CLINICAL TRIAL: NCT07017998
Title: Mild Therapeutic Hypothermia for Tinnitus Management
Brief Title: External Therapy for Tinnitus Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Restorear Devices LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-FY2025-39
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Tinnitus; Tinnitus, Subjective
Keywords: tinnitus; ringing in the ears; ringing ears; symptom management; cooling; red light therapy
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: The study is a prospective, single-blind and decentralized randomized control study. All study procedures and data collection will be completed by participants remotely using online modules under the guidance of an audiologist.
  Participants will be sent a test kit to complete the study procedures on their own time and will access an online module for data collection via Qualtrics XM. Participants will be asked to use a wearable, headband-style device and to respond to questions about their tinnitus experience.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Experimental Arm (Experimental): Participants will wear a headband-style device for 30 minutes in a single session. Subjective assessments will be completed via Qualtrics XM, and responses will be compared to those in the Sham Arm. n=40
  Interventions: Device: Cold pack-delivered mild therapeutic hypothermia
- Control Arm (Sham Comparator): Participants will wear a headband-style control device for a single 30 minute session. Subjective assessments will be completed via Qualtrics XM, and responses will be compared to those in the Experimental Arm. n=40
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: Cold pack-delivered mild therapeutic hypothermia — Mild therapeutic hypothermia (cooling), delivered non-invasively to the structures of the inner ear (cochlea) for 30 minutes, using headband-style proprietary device, ReBound.
  Arms: Experimental Arm
Device: Sham (No Treatment) — Sham headband-style device will be worn for 30 minutes. Participants will be told they are receiving therapy.
  Arms: Control Arm

SUMMARY:
The goal of this remote interventional clinical study is to investigate the use of mild therapeutic hypothermia devices for the symptomatic relief of chronic tinnitus. The main aims of the study are:

1. Ascertain the effects of MTH in chronic tinnitus patients using questionnaires measuring tinnitus severity and intervention-related change.
2. Ascertain the comfort and acceptability of the hypothermia device and therapy.

Participants with chronic tinnitus will wear the mild therapeutic hypothermia therapy devices for a single 30 minute session. Researchers will compare results from those receiving therapy to those from a control group.

DETAILED DESCRIPTION:
Tinnitus is the perception of sound in the absence of an external stimulus, commonly described as ringing in the ears. Tinnitus is a highly common condition, with most individuals experiencing it at some point in their lifetime. At least 1 in 10 US adults experience chronic or disabling tinnitus, with a significant negative impact on quality of life, often affecting sleep, concentration, mood, and hearing ability. Tinnitus can be intermittent or constant in nature, and intensity can vary or be exacerbated by stress, noise exposure, or other factors. Currently, there is no widely applicable cure for tinnitus, and management typically includes use of sound therapy, mental health counseling, lifestyle modifications, stress management, and distraction techniques. Tinnitus is associated with changes in auditory function, with hearing loss being the most commonly associated co-morbidity in patients. However, tinnitus can also be observed in patients with normal hearing.

Tinnitus can have a significant deleterious effect on a person's quality of life, and there is currently no cure. State-of-the art treatment options suffer limitations and are often ineffective and complex. Most widely used tinnitus treatments focus on reducing awareness of tinnitus/masking symptoms and the impact on emotional state rather than seeking to address the underlying mechanisms of the sound generation. Treatment modalities include sound therapy using environmental sounds and/or hearing aids, psychological interventions including tinnitus retraining therapy and/or cognitive behavioral therapy, somatosensory stimulation including vagus nerve stimulation and osteopathic manipulation, and distraction exercises including guided breathing and development of new hobbies. Other therapies aim to target the generation of tinnitus, including direct and indirect stimulation of the auditory cortex and/or other brain structures through neuromodulation and pharmacologic intervention. Despite the limited success of many of these treatment modalities, none have been shown to be widely applicable to manage tinnitus severity or provide a treatment for tinnitus.

Modifying temperature of the cochlea is known to influence auditory responses. The study team and others have shown that MTH delivered locally or systemically protects hearing function and cochlear structures against noise-induced hearing loss when compared to normothermic animals. It has also been shown in preclinical studies that MTH is safe. Lamprecht and Morgenstern first observed changes in tinnitus intensity in response to warm and cool caloric irrigations, and they found irrigation with warm (44ºC) water was associated with a perceptual increase in tinnitus, while irrigation with cool (30ºC) water was associated with a perceptual decrease in tinnitus. Recently, the idea of using cool water irrigation to reduce tinnitus was further explored. They found that irrigation with cool water resulted in a decrease in tinnitus perception as well as tinnitus disturbance as measured by the Tinnitus Handicap Inventory (THI).

In this study, investigators aim to show the efficacy of a highly accessible and translatable, non-invasive treatment strategy and device utilizing mild therapeutic hypothermia, or MTH, to reduce tinnitus symptom severity in patients with chronic tinnitus. The study team has designed and manufactured the headband-style device, ReBound, to provide therapeutic hypothermia to the inner ear structures. The aims of the study are:

Aim 1: Ascertain the effects of MTH in chronic tinnitus patients using questionnaires measuring tinnitus severity and intervention-related change. After collection of validated subjective assessments (adapted tinnitus Visual Analog Scale (VAS)) MTH will be delivered bilaterally for 30 minutes in a home setting using custom cold packs placed securely on the temporal bone. Half of the participants will receive a placebo treatment via sham devices. Pre- and post-assessments will be compared between normothermic (sham) and MTH-treated patients at completion of treatment and 24-hours post-treatment. Any adverse events (caloric activation of the vestibular system, skin frostbite) will be closely monitored by an audiologist. Results of Aim 1 will establish MTH as a novel approach for tinnitus symptom management.

Aim 2: Ascertain the comfort and acceptability of the device and therapy. Participants will be given a 6-question Device Acceptance Questionnaire (DAQ) in their post-assessment detailing their subjective experience of the comfort and acceptability of the therapy. They will rate their experience with the ease of use, comfort, and overall satisfaction with the device on a scale of 1-4.

This study will be completed entirely remotely and asynchronously in participants' homes. This research will be highly impactful given the significant adverse effects of tinnitus, an unmet clinical need, and the high translational potential of MTH for managing tinnitus severity.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-55 years of age at the time of signing the informed consent form with primary complaint of tinnitus;
* Suffering from subjective tinnitus for at least 30 days;
* Tinnitus whose level of severity is defined by Tinnitus Handicap Inventory (THI) values ≥12,
* Tinnitus is constant in nature (defined as audible at least 75% of waking hours).

Exclusion Criteria:

* Very mild tinnitus (THI values <12);
* Tinnitus that is intermittent in nature;
* Tinnitus described as non-auditory or pulsatile in nature;
* Individuals with a history of vertigo or fluctuating hearing loss, such as that related to Menière's disease, chronic otitis, vestibular neuritis, neuroma, otosclerosis cholesteatoma, or temporomandibular joint disorder;
* Individuals with a history of extreme sensitivity to cold or heat, including individuals with a past history of frostbite or Raynaud's Syndrome.
* Those who are currently receiving medical, pharmacologic, or therapeutic intervention for tinnitus or other otologic conditions, including sound therapy, cognitive behavioral therapy (CBT), Tinnitus Retraining Therapy (TRT), steroid injections, or other treatments;
* Those who present with a mental health score indicating significant psychological component, per standard of care, based on PHQ-4 score of moderate to severe anxiety/depression.
* Children (under 18 years), incarcerated individuals, adults unable to consent, and psychologically vulnerable participants.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Subjective Tinnitus Severity | Immediately prior to and immediately after treatment or sham treatment.
  An adapted 4-question visual analog scale (VAS) will be used to assess tinnitus awareness, loudness, tolerance and disturbance before baseline treatment and repeated immediately after application using the online survey module. The VAS has been adapted to address the current, acute subjective experience of the participants' tinnitus rather than their general experience. The VAS consists of a sliding scale from 0 to 100, with 100 correlating to a greater disease burden/worse symptoms.

SECONDARY OUTCOMES:
Perceived Improvement of Tinnitus Symptoms | Immediately after treatment or sham treatment.
  The Patient Global Impression of Improvement (PGI-I) scale will be administered immediately post-treatment using the online survey module. This scale will allow participants to rank, subjectively, how their tinnitus compares after treatment versus to before. The PGI-I is a written rather than numerical scale, with potential values ranging from "very much better" to "very much worse".
Comfort and Acceptability Questionnaire | Immediately after treatment in the Experimental Arm.
  A 6-item Device Acceptance Questionnaire (DAQ) will be used to assess the comfort and acceptability of the therapy (Aim 2). DAQ will be administered immediately after treatment in the experimental group. The DAQ consists of Likert scale questions pertaining to the comfort of the device, with responses including: "strongly disagree", "disagree", "agree", and "strongly agree".
Adverse Events Questionnaire | Immediately after treatment or sham treatment.
  A 2-question Adverse Event Questionnaire (AEQ) will be administered immediately post-treatment to record any mild adverse events associated with the therapy, including headache, dizziness, or irritation. Participants will identify adverse events they experienced from a provided list, with the option to add their own.

CONTACTS AND LOCATIONS:
Overall Officials: Suhrud Rajguru, PhD, Principal Investigator — RestorEar Devices; Kendall Stern, MPH, Principal Investigator — RestorEar Devices
Locations (1):
- RestorEar Devices, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saatci, O., O.A. Duz, and N.G.Y. Aslier, Efficacy of caloric vestibular stimulation for the treatment of idiopathic tinnitus. Journal of Surgery and Medicine, 2020. 4(11): p. 1041-1045.
- [Background] Lamprecht J, Morgenstern C. [Bilateral caloric long-term irrigation as a method for the differentiation of tonal tinnitus]. Laryngol Rhinol Otol (Stuttg). 1985 Jan;64(1):17-20. German. PMID 3968937
- [Background] Rincon Sabatino S, Rivero A, Sangaletti R, Dietrich WD, Hoffer ME, King CS, Rajguru SM. Targeted therapeutic hypothermia protects against noise induced hearing loss. Front Neurosci. 2024 Jan 16;17:1296458. doi: 10.3389/fnins.2023.1296458. eCollection 2023. PMID 38292902
- [Background] Rincon Sabatino S, Sangaletti R, Griswold A, Dietrich WD, King CS, Rajguru SM. Transcriptional response to mild therapeutic hypothermia in noise-induced cochlear injury. Front Neurosci. 2024 Jan 17;17:1296475. doi: 10.3389/fnins.2023.1296475. eCollection 2023. PMID 38298897
- [Background] Tamames I, King C, Huang CY, Telischi FF, Hoffer ME, Rajguru SM. Theoretical Evaluation and Experimental Validation of Localized Therapeutic Hypothermia Application to Preserve Residual Hearing After Cochlear Implantation. Ear Hear. 2018 Jul/Aug;39(4):712-719. doi: 10.1097/AUD.0000000000000529. PMID 29240567
- [Background] Tamames I, King C, Bas E, Dietrich WD, Telischi F, Rajguru SM. A cool approach to reducing electrode-induced trauma: Localized therapeutic hypothermia conserves residual hearing in cochlear implantation. Hear Res. 2016 Sep;339:32-9. doi: 10.1016/j.heares.2016.05.015. Epub 2016 May 31. PMID 27260269
- [Background] Henry KR. Hyperthermia exacerbates and hypothermia protects from noise-induced threshold elevation of the cochlear nerve envelope response in the C57BL/6J mouse. Hear Res. 2003 May;179(1-2):88-96. doi: 10.1016/s0378-5955(03)00097-2. PMID 12742241
- [Background] Watanabe F, Koga K, Hakuba N, Gyo K. Hypothermia prevents hearing loss and progressive hair cell loss after transient cochlear ischemia in gerbils. Neuroscience. 2001;102(3):639-45. doi: 10.1016/s0306-4522(00)00510-8. PMID 11226700
- [Background] Henry KR, Chole RA. Hypothermia protects the cochlea from noise damage. Hear Res. 1984 Dec;16(3):225-30. doi: 10.1016/0378-5955(84)90111-4. PMID 6401081
- [Background] Meisel-Mikolajczyk F, Swoboda-Kopec E, Skoskiewicz M. [Isolation of Bacteroides fragilis from the appendix in a case of appendicitis]. Pol Tyg Lek. 1977 Aug 1;32(31):1209-10. No abstract available. Polish. PMID 896576
- [Background] Liberman MC, Dodds LW. Single-neuron labeling and chronic cochlear pathology. II. Stereocilia damage and alterations of spontaneous discharge rates. Hear Res. 1984 Oct;16(1):43-53. doi: 10.1016/0378-5955(84)90024-8. PMID 6511672
- [Background] Brown MC, Smith DI, Nuttall AL. The temperature dependency of neural and hair cell responses evoked by high frequencies. J Acoust Soc Am. 1983 May;73(5):1662-70. doi: 10.1121/1.389387. PMID 6863743
- [Background] Eggermont JJ, Roberts LE. The neuroscience of tinnitus: understanding abnormal and normal auditory perception. Front Syst Neurosci. 2012 Jul 11;6:53. doi: 10.3389/fnsys.2012.00053. eCollection 2012. No abstract available. PMID 22798948
- [Background] Sheldrake J, Diehl PU, Schaette R. Audiometric characteristics of hyperacusis patients. Front Neurol. 2015 May 15;6:105. doi: 10.3389/fneur.2015.00105. eCollection 2015. PMID 26029161
- [Background] Sanchez TG, Medeiros IR, Levy CP, Ramalho Jda R, Bento RF. Tinnitus in normally hearing patients: clinical aspects and repercussions. Braz J Otorhinolaryngol. 2005 Jul-Aug;71(4):427-31. doi: 10.1016/s1808-8694(15)31194-0. Epub 2005 Dec 15. PMID 16446955
- [Background] Baguley D, McFerran D, Hall D. Tinnitus. Lancet. 2013 Nov 9;382(9904):1600-7. doi: 10.1016/S0140-6736(13)60142-7. Epub 2013 Jul 2. PMID 23827090